CLINICAL TRIAL: NCT05289882
Title: Purpose After Service Through Sport (PASS)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit sufficient sample to commence trial
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Mark Beauchamp, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H21-02693
Record Dates: First submitted 2022-03-03; First posted 2022-03-22 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Well-Being (Psychological Flourishing)
Keywords: Mental Health; Physical Health; Military Veterans; Social Connectedness; Men's Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Using Optimal Design Software, and on the basis of 7 observations per participant (in psychological flourishing), 134 participants are required to detect a medium effect size of δ = .50, with Power (1 - β) set at 80%, and p <.05 with seven time points (baseline, Months 1, 2, 3, 4, 5, and 6). To account for 9 sites across Canada (necessitating 8 dummy variables) requires an additional 80 participants. To further account for 10% attrition, a minimum of n= 238 veteran participants are needed. The study will look to recruit 252 military veterans for study participation. The study will also look to recruit N = 252 currently serving members of the Canadian Armed Forces, although it should be noted that these participants do not constitute the population of primary interest for the trial. On the basis of N = 252 military veterans and N = 252 currently serving military participants the trial will look to recruit a total of N = 504 participants.
Who Masked: Outcomes Assessor
Masking Description: Personnel who analyze the data collected from the study are not aware of the treatment applied to any given group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PASS Program Condition (Experimental): Participants in this condition will take part in weekly physical activity, augmented with built-in opportunities to socially connect, and be directed to veteran-specific support services and resources.
  Interventions: Behavioral: PASS Program Condition:
- Waitlist Control (No Intervention): Those randomized to the wait-list control condition will go about their daily lives for the duration of the 6-month assessment period (following randomization). They will be asked to complete the same measures (and will be remunerated in the same way as those in the PASS program condition, based on the completion of study measures). At the end of the 6-month trial, participants in this condition will have the opportunity to participate in the PASS program.

INTERVENTIONS:
Behavioral: PASS Program Condition: — Participants randomized to this condition will be invited to take part in weekly ball hockey games (once per week), that will last approximately 60 minutes, and will be followed by opportunities to socially connect afterwards. The results of our feasibility study indicated that the PASS program acted as an important conduit to direct participants to other support services and resources (e.g., counseling, career transition centre, employment, education). Military veteran men are often reluctant to access such supports, especially if they attach stigma to such services (e.g., mental health services). At each site, a military veteran will be trained as a facilitator to operate as a conduit to refer participants to the relevant support services and agencies.
  Arms: PASS Program Condition

SUMMARY:
The purpose of this study is to evaluate the efficacy of a gender-sensitized social-connectedness physical activity program in relation to key markers of well-being among military veteran men over 6 months.

DETAILED DESCRIPTION:
The transition to civilian life can bring about substantive challenges for military veterans. Particular challenges include a loss of identity, feelings of loneliness and isolation, difficulties with finding and retaining employment, substance misuse, and problems adjusting to very different work and cultural environments. A growing body of scientific evidence also indicates that military veterans are at notable risk of depleted mental health (e.g., depression, suicide ideation).

The study involves broadening the evaluation (e.g., assess its impact on mental and physical health) and reach (e.g. extend to other Canadian cities) of a recently developed pilot program, Purpose After Service through Sport (PASS), which was completed in Vancouver in 2020 and assessed for its feasibility and acceptability. The results from this pilot study revealed that the program was well-received (by both military leadership and veterans themselves), fostered a sense of social connectivity among veterans, resulted in (self-reported) physical and psychological health benefits, and displayed considerable potential for scale up and evaluation using a randomized controlled trial (RCT) design.

The PASS Randomized Trial draws from the empirical evidence related to (a) the mental health benefits of regular physical activity, (b) benefits of group-based programs that foster social connectivity, (c) the importance of, and potential derived from, developing and implementing gender-sensitized programs, and (d) the pilot study described above.

ELIGIBILITY:
Inclusion Criteria:

* Former members of the Canadian (or Allied Forces; e.g., NATO countries) military, or current members of the Canadian military, and not experience any contraindication which might prevent that person from participating in moderate-intensity physical activity.
* Self-identification as a man (if sex at birth is 'female' but participants identify as 'man' they are eligible to participate).
* Have received full dosage of the COVID-19 vaccination (min 2 injections) and must provide proof of vaccination, as this is required to access all active military bases in Canada.
* Be able to read and understand English or French.
* Have access to a computer, tablet, or other device, that has access to the internet.
* Live at, or in close proximity to, one of the nine study locations (Esquimalt, BC; Edmonton, AB, Shilo, MB; Borden, ON; Kingston, ON; Petawawa, ON; Valcartier, QC; Montreal, QC; Gagetown, NB)

Exclusion Criteria:

* Not a former member of the Canadian (or Allied Forces; e.g., NATO countries) military, or current member of the Canadian military.
* Unable to participate in moderate-intensity physical activity (as screened via the PAR-Q and ePARmedX), including a lack of ability to receive doctor's clearance for participating in physical activity.
* Unable to speak or read English or French
* Lack of internet access which prevents access to online materials (e.g., questionnaires).
* Participants do not self-identify as 'man'. If participants disclose 'sex' as female but self-identify their gender identity as 'man' they are eligible to participate in the study and we would include their psychological responses in the main analyses. In such an instance, their biological measures (blood draws, blood pressure, and physical fitness tests) would be analyzed separately from those whose sex (male) and gender identity (man) are concordant.
* Not living in proximity to one of the participating sites (in order to take part in the in-person group-based activities).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Self-identification as a man
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in well-being (psychological flourishing) over the course of the intervention | Tracked monthly for 6 months (baseline, followed by 6 months of intervention)
  Diener's (2010) flourishing scale will be used in the baseline survey, and will be in each monthly survey to track changes in flourishing over the study period. There are 8 items, phrased in a positive direction. Scores can range from 8 (strong disagreement with all items) to 56 (strong agreement with all items), with higher scores indicating individuals who have a more positive view of themselves in important areas of functioning.

SECONDARY OUTCOMES:
Changes in life satisfaction over the course of the intervention | Tracked monthly for 6 months (baseline, followed by 6 months of intervention)
  Life satisfaction will be assessed using the 1-item question by Fleeson (2004), with responses anchored from 0 to 10 where 0 means "the worst possible life overall" and 10 means "the best possible life overall".
Change in global physical and mental health over the course of the intervention | Tracked monthly for 6 months (baseline, followed by 6 months of intervention)
  Global indicators of physical and mental health will be assessed using items by Hays et al. (2009), each anchored on a 5-point scale (1 = "poor", 5 = "excellent") with higher scores reflecting better physical and mental health.
Change in stress over the course of the intervention | Tracked monthly for 6 months (baseline, followed by 6 months of intervention)
  The 1-item Statistics Canada (2012) stress question will be used in the baseline survey and in monthly surveys to track changes in psychological stress over the study period. The SCSQ is a 1-item question, with responses anchored on a 5-point scale, with a possible scoring of 1 ("not at all stressful") to 5 ("extremely stressful"), with higher scores indicating more stress.
Change in anxiety over the course of the intervention | Tracked monthly for 6 months (baseline, followed by 6 months of intervention)
  The 7-item generalized anxiety disorder scale (Spitzer et al., 2006) will be used to assess anxiety symptoms. Items are anchored on a 4-point scale (0 = "not at all" to 3 = "nearly every day") with higher scores indicative of more frequent experience of anxiety symptoms.
Change in post-traumatic stress disorder symptomology over the course of the intervention | Tracked monthly for 6 months (baseline, followed by 6 months of intervention)
  The 20-item PTSD checklist for diagnostic and statistical manual of mental disorders-fifth edition (Bovin, 2016) will be used to assess PTSD symtomology. Items are anchored on a 5-point scale (1 = "not at all", 5 = "extremely") with higher scores reflective of higher levels of PTSD symptomology.
Change in depression over the course of the intervention | Tracked monthly for 6 months (baseline, followed by 6 months of intervention)
  The 10-item center for epidemiologic studies depression scale by Andresen et al. (1994) will be used in the baseline survey, and will be in each monthly survey to track changes in depression symptoms over the study period. The possible range in scores is 0 to 30 depending on number of symptoms, with those symptoms weighted by frequency experienced in a week. Higher scores indicate more or more frequent symptoms.
Change in resilience over the course of the intervention | Tracked monthly for 6 months (baseline, followed by 6 months of intervention)
  The brief resilience scale by Smith et al. (2008) will be used in the baseline survey, and will be in each monthly survey to track changes in resilience over the study period. This instrument uses a mean scoring system with a possible range in scores from 1-5; higher scores indicate the individual perceives they have a better ability to 'bounce back' and recover from stressful events and/or situations.
Change in social identification over the course of the intervention | Tracked monthly for 6 months (baseline, followed by 6 months of intervention)
  The degree to which participants in the intervention condition identify with others in the program will be assessed using items adapted from the 4-item scale by Doosje et al. (1995). Note that this measure will only be administered to participants in the experimental (i.e., intervention) condition. Items are anchored on a 7-point scale (1 = "strongly disagree", 7 = "strongly agree") with higher scores reflecting greater social identification with the group.
Change in social connectedness over the course of the intervention | Tracked monthly for 6 months (baseline, followed by 6 months of intervention)
  Social connectedness will be assessed using the 20-item social connectedness scale - revised (Lee et al., 2001). Items are anchored on a 6-point scale (1 = "strongly disagree", 6 = "strongly agree") with higher scores reflecting greater social connectedness with others.
Change in loneliness over the course of the intervention | Tracked monthly for 6 months (baseline, followed by 6 months of intervention)
  Loneliness will be assessed using the 3-item loneliness scale (Hughes et al., 2004) in which items are anchored on a 3-point scale (1 = "hardly ever", 3 = "often") with higher scores reflecting greater loneliness.
Change in leisure-time physical activity over the course of the intervention | Tracked monthly for 6 months (baseline, followed by 6 months of intervention)
  Leisure-time physical activity will be assessed using a modified version of the leisure score index (Courneya et al, 2004) that has been applied to Godin's leisure time exercise questionnaire (Godin & Shepard, 1985). Participants report the frequency per week and time per exercise session of any mild, moderate, or strenuous exercise that participants complete.
Change in sleep quality over the course of the intervention | Tracked monthly for 6 months (baseline, followed by 6 months of intervention)
  Sleep quality will be assessed using the 1-item measure developed by Buysse et al. (1989), that is anchored on a 4-point scale (1 = "very bad", 4 = "very good") with higher scores reflective of better sleep.
Program adherence over the course of the intervention | Weekly attendance at PASS program sessions over 6 month intervention
  Assessed using program logs maintained by location managers (intervention condition only).
Access and use of health services over the course of the intervention | Assessed over 6 months (descriptive measure)
  Assessed, among intervention participants only, with a single question, "As a result of the PASS program, have you accessed support services for any of the following areas of need?", followed by an indication of which services were accessed, if any.

OTHER OUTCOMES:
Physical fitness | Baseline (Month 0) and 6-month post PASS program commencement
  Assessed using the multistage fitness test (Leger & Lambert, 1982). There are 21 possible levels, with higher scores indicating better fitness.
HbA1c | Baseline (Month 0) and 6-month post PASS program commencement
  A hemoglobin A1c (HbA1c) test measures the amount of blood sugar (glucose) attached to hemoglobin. Higher levels of HbA1c are indicative of higher levels of circulating glucose levels.
Systolic and Diastolic Blood Pressure. | Baseline (Month 0) and 6-month post PASS program commencement
  Assessed using a standard sphygmomanometer. Blood pressure of less than 120/80 mm Hg is considered within the normal range. Elevated blood pressure exists when readings range from 120-129 systolic and less than 80 mm Hg diastolic. Hypertension Stage 1 exists when blood pressure ranges from 130-139 systolic or 80-89 mm Hg diastolic. Hypertension Stage 2 exists when blood pressure exists at 140/90 mm Hg or higher. A Hypertensive Crisis (requires medical attention) exists if blood pressure exceeds 180/120 mm Hg.
C-reactive Protein (CRP) | Baseline (Month 0) and 6-month post PASS program commencement
  C-reactive protein (CRP) provides an indication of inflammation in the body. Higher levels of CRP are indicative of greater inflammation.
Telomere Length | Baseline (Month 0) and 6-month post PASS program commencement
  Telomere length provides an indication of cell aging, and is assessed using a polymerase chain reaction (PCR) test. Shorter telomeres indicate greater cell aging.

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Beauchamp, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
The protocol for the study is available on the Open Science Framework (embargoed until 31/10/2022, to allow for study completion). The statistical analysis plan is also available on the Open Science Framework (embargoed until 31/10/2022). The consent form is freely available if requested from the Primary Investigator (Beauchamp, M).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available from this trial 1 year after completion of the study. The data will remain available indefinitely.
Access Criteria: The nature of the request for sharing access will be reviewed by the PI (Beauchamp, M) and the data management team. Data will be shared via secure platforms (Redcap). Contact for data access can be done through personal communication (e.g., email) with PI Beauchamp (mark.beauchamp@ubc.ca).

REFERENCES:
- [Background] Andresen EM, Malmgren JA, Carter WB, Patrick DL. Screening for depression in well older adults: evaluation of a short form of the CES-D (Center for Epidemiologic Studies Depression Scale). Am J Prev Med. 1994 Mar-Apr;10(2):77-84. PMID 8037935
- [Background] Bovin MJ, Marx BP, Weathers FW, Gallagher MW, Rodriguez P, Schnurr PP, Keane TM. Psychometric properties of the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (PCL-5) in veterans. Psychol Assess. 2016 Nov;28(11):1379-1391. doi: 10.1037/pas0000254. Epub 2015 Dec 14. PMID 26653052
- [Background] Courneya KS, Jones LW, Rhodes RE, Blanchard CM. Effects of different combinations of intensity categories on self-reported exercise. Res Q Exerc Sport. 2004 Dec;75(4):429-33. doi: 10.1080/02701367.2004.10609176. No abstract available. PMID 15673042
- [Background] Dallaire RA, Wells DM. The transition to civilian life of veterans. 2014. www.senate-senat.ca/veac.asp
- [Background] Diener E, Wirtz D, Biswas-Diener R, Tov W, Kim-Prieto C, Choi D-W, Oishi S. New measures of well-being: Short scales to assess flourishing and positive and negative feelings. Soc Indic Res. 2010;97, 143-156.
- [Background] Doosje B, Ellemers N, Spears R. Perceived intragroup variability as a function of group status and identification. J Exp Soc Psychol. 1995;31(5), 410-436.
- [Background] Feingold A. New Approaches for Estimation of Effect Sizes and their Confidence Intervals for Treatment Effects from Randomized Controlled Trials. Quant Method Psychol. 2019;15(2):96-111. doi: 10.20982/tqmp.15.2.p096. PMID 32775313
- [Background] Feingold A. Effect sizes for growth-modeling analysis for controlled clinical trials in the same metric as for classical analysis. Psychol Methods. 2009 Mar;14(1):43-53. doi: 10.1037/a0014699. PMID 19271847
- [Background] Feingold A. A Regression Framework for Effect Size Assessments in Longitudinal Modeling of Group Differences. Rev Gen Psychol. 2013 Mar;17(1):111-121. doi: 10.1037/a0030048. PMID 23956615
- [Background] Fleeson W. The quality of American life at the end of the century. In Brim OG, Ryff CD, Kessler RC (Eds.), How healthy are we?: A national study of well-being at midlife. 2004. University of Chicago Press.
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Hays RD, Bjorner JB, Revicki DA, Spritzer KL, Cella D. Development of physical and mental health summary scores from the patient-reported outcomes measurement information system (PROMIS) global items. Qual Life Res. 2009 Sep;18(7):873-80. doi: 10.1007/s11136-009-9496-9. Epub 2009 Jun 19. PMID 19543809
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- [Background] Kvam S, Kleppe CL, Nordhus IH, Hovland A. Exercise as a treatment for depression: A meta-analysis. J Affect Disord. 2016 Sep 15;202:67-86. doi: 10.1016/j.jad.2016.03.063. Epub 2016 May 20. PMID 27253219
- [Background] Lee RM, Draper M, Lee S. Social connectedness, dysfunctional interpersonal behaviors, and psychological distress: Testing a mediator model. J Couns Psychol. 2001; 48(3), 310-318.
- [Background] Leger LA, Lambert J. A maximal multistage 20-m shuttle run test to predict VO2 max. Eur J Appl Physiol Occup Physiol. 1982;49(1):1-12. doi: 10.1007/BF00428958. PMID 7201922
- [Background] McCreary, D. R. (2019). Veteran and first responder mental il health and suicide prevention: A scoping review of prevention and early intervention programs used in Canada, Australia, New Zealand, Ireland, and the United Kingdom. British Columbia, Canada: Donald McCreary Scientific Consulting.
- [Background] McDowell CP, Dishman RK, Gordon BR, Herring MP. Physical Activity and Anxiety: A Systematic Review and Meta-analysis of Prospective Cohort Studies. Am J Prev Med. 2019 Oct;57(4):545-556. doi: 10.1016/j.amepre.2019.05.012. PMID 31542132
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Background] Raudenbush SW, Spybrook J, Congdon R, Liu X, Martinez A. Optimal Design Software for Multi-level and Longitudinal Research (Version 2.01) [Software]. 2011. www.wtgrantfoundation.org
- [Background] Rosenbaum S, Vancampfort D, Steel Z, Newby J, Ward PB, Stubbs B. Physical activity in the treatment of Post-traumatic stress disorder: A systematic review and meta-analysis. Psychiatry Res. 2015 Dec 15;230(2):130-6. doi: 10.1016/j.psychres.2015.10.017. Epub 2015 Oct 20. PMID 26500072
- [Background] Shields DM, Kuhl D, Lutz K, Frender J, Baumann, N., Lopresti P. Mental health and well-being of military veterans during military to civilian transition: Review and analysis of the recent literature. 2016. https://doi.org/10.13140/RG.2.2.14092.62084
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Statistics Canada. (2012). Canadian Community Health Survey (CCHS) - Mental Health. http://www23.statcan.gc.ca/imdb/p2SV.pl?Function=getSurvey&SDDS=5015#a2
- [Background] Steffens NK, LaRue CJ, Haslam C, Walter ZC, Cruwys T, Munt KA, Haslam SA, Jetten J, Tarrant M. Social identification-building interventions to improve health: a systematic review and meta-analysis. Health Psychol Rev. 2021 Mar;15(1):85-112. doi: 10.1080/17437199.2019.1669481. Epub 2019 Oct 7. PMID 31530154
- [Background] Tam CC, Zeng C, Li X. Prescription opioid misuse and its correlates among veterans and military in the United States: A systematic literature review. Drug Alcohol Depend. 2020 Nov 1;216:108311. doi: 10.1016/j.drugalcdep.2020.108311. Epub 2020 Sep 21. PMID 33010713
- [Background] Waldhauser KJ, O'Rourke JJ, Jackson B, Dimmock, JA, Beauchamp MR. Purpose after service through sport: A social identity-informed program to support military veteran well-being. Sport Exerc Perform Psychol. 2021;10(3), 423-437.
- [Background] Wilson G, Hill M, Kiernan MD. Loneliness and social isolation of military veterans: systematic narrative review. Occup Med (Lond). 2018 Dec 26;68(9):600-609. doi: 10.1093/occmed/kqy160. PMID 30551163